CLINICAL TRIAL: NCT06233747
Title: I-CARE: The Effectiveness of a Modular Digital Intervention to Reduce Suicidal Ideation and Emotional Distress During Pediatric Psychiatric Boarding
Brief Title: Improving Care, Accelerating Recovery and Education
Acronym: I-CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Dartmouth College (Other); Children's Hospital of Philadelphia (Other); University of Vermont (Other)
Responsible Party: Principal Investigator, JoAnna K. Leyenaar, Principal Investigator; Staff Physician; Professor of Pediatrics, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02002045; RF1MH134626 (NIH)
Record Dates: First submitted 2024-01-12; First posted 2024-01-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Disorder; Suicide Attempt; Suicidal Ideation; Emergency Psychiatric
Keywords: children; adolescents; emergency department; psychosocial skills; mental health boarding
MeSH Terms: conditions — Mental Disorders; Suicide, Attempted; Suicidal Ideation; Emergencies | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge pilot study, in which 2 hospitals will be randomized to begin implementation of I-CARE at 2 different times within the 17-month study period. Both sites begin with an initial 3-month period of treatment-as-usual and the research team collects all outcome measures during this period, then 1 hospital will crossover to launch the I-CARE intervention and the other will launch 2 months later (continuing to provide treatment-as-usual in the interim). This may be considered a form of a parallel cluster study, in which one of the two hospitals is initially randomized to I-CARE while the other remains in the baseline/treatment-as-usual state.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-CARE (Experimental): I-CARE (Improving Care, Accelerating Recovery & Education) is a quality improvement program designed to deliver evidence-based psychosocial skills to adolescents during mental health boarding. The program consists of 7 web-based animated videos and workbook exercises, facilitated by licensed nursing assistants/behavioral health technicians/safety attendants who provide one-on-one safety supervision during boarding. I-CARE will be offered to all eligible adolescents who are boarding and only those who agree to participate in a program evaluation will be involved in the research component.
  Interventions: Behavioral: Improving Care, Accelerating Recovery & Education (ICARE)
- Usual Care (No Intervention): These hospitals currently offer basic safety supervision and medical monitoring for adolescents during mental health boarding. This is the "usual care" condition.

INTERVENTIONS:
Behavioral: Improving Care, Accelerating Recovery & Education (ICARE) — I-CARE is a brief, digital intervention designed for adolescents who are boarding in a medical hospital awaiting transfer to a psychiatric inpatient unit. It consists of 7 tablet-based animated video modules and workbook exercises, facilitated by licensed nursing assistants or other non-specialist clinicians who provide one-on-one safety supervision during boarding. All modules are grounded in evidence-based practices, such as cognitive-behavioral therapy and dialectical behavior therapy. Given that one-on-one safety supervision is the current standard of care during boarding, I-CARE requires minimal additional resources beyond those already available in acute care hospitals and builds on well established research demonstrating the effectiveness of task-sharing, the redistribution of tasks within the workforce, to address the shortage of mental health professionals.
  Arms: I-CARE

SUMMARY:
The goal of this clinical trial is to test the I-CARE program in children who are in a medical hospital awaiting inpatient mental health treatment. The main questions it aims to answer are:

* Can the I-CARE program be used at the medical hospitals and do the patients and hospital staff like the program?
* Does the I-CARE program lower patients' emotional distress, thoughts about suicide or suicide attempts?

Patients will complete as many of the 7 I-CARE videos as possible during their stay at the medical hospital and fill out online surveys. There are workbook activities that go with each I-CARE video. A hospital staff member will help the patient do the videos and workbook activities.

DETAILED DESCRIPTION:
The COVID-19 pandemic has contributed to a dramatic and unprecedented rise in pediatric mental health conditions, with rates of depression and anxiety doubling from pre-pandemic estimates. These increases exacerbate decades-long trends of increasing youth suicidality. Suicide is the second leading cause of death among adolescents; from 2007 to 2017 suicide deaths tripled in youth 10 to 14 years. Emergency departments (EDs) at acute care hospitals increasingly serve as portals of care for youth with suicidal ideation or attempt. When these youth are deemed to require psychiatric hospitalization, the demand for beds often exceeds supply, leading to psychiatric boarding. To address this gap, a multidisciplinary team including pediatricians, psychologists and patient partners developed a modular digital intervention and associated training materials to deliver evidence-based psychosocial skills to youth during boarding. This program, entitled I-CARE (Improving Care, Accelerating Recovery & Education), consists of 7 web-based animated videos and workbook exercises, facilitated by licensed nursing assistants who provide 1-on-1 safety supervision during boarding. Given that 1-on-1 safety supervision is the current standard of care at most hospitals, I-CARE requires minimal additional resources beyond those already available in these settings. The psychosocial skills included in I-CARE are grounded in cognitive behavioral therapy and were prioritized through a rigorous Delphi process evaluating their importance and feasibility to deliver during psychiatric boarding.

Aim 1:

Adapt and refine I-CARE training and implementation materials, taking into account variation in hospital resources and boarding locations while maintaining implementation fidelity.

Aim 2:

Using an open pilot/case series design, assess I-CARE feasibility and engagement of target mechanisms from the perspectives of youth, caregivers, and clinicians using a mixed-methods approach.

Aim 3:

Determine the preliminary effectiveness of I-CARE to reduce emotional distress and suicidal risk compared to usual care in youth experiencing boarding for suicidal ideation or attempt, and assess the effects of I-CARE on readiness for change, suicide-related coping, hope, and mental health treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-17 years
* Ability to speak and complete surveys in English
* Presented to ED with suicidal ideation or attempt
* Awaiting psychiatric disposition
* Receiving one-on-one safety supervision
* Medically stable

Exclusion Criteria:

* Cognitive or developmental delays that preclude program participation based on clinical team assessment
* Diagnosis of psychosis
* Primary reason for hospitalization or ED visit is an eating disorder
* Parent/guardian not able to provide consent in English
* Admission or transfer for psychiatric care anticipated on the first day of potential enrollment
* Clinical team concern for patient or staff safety based upon active behavioral concerns
* In child protective custody/ward of the state

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depression, Anxiety, and Stress Scale, Youth (DASS-Y) | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 3 months (T4), and 6 months (T5) post-discharge
  The DASS-Y is a 21-item, youth-oriented validated measure that generates an aggregate assessment of emotional distress and sub-measures of depression, anxiety, and stress. Each item is self-reported on a 4-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much, or most of the time).
Change in Harkavy-Asnis Suicide Scale (HASS), Suicide Attempt Module (HASS) | 30 days (T3), 3 months (T4), and 6 months (T5) postdischarge
  The HASS consists of 21 self-report items that cover the range of suicidal ideation and attempts, including both passive and active ideation. Responses on each item range 0-4; total scores range 0-84, with higher scores indicating more severe suicidality. The study will use only the 2 questions that inquire about suicide attempts.
Change in Concise Health Risk Tracking (CHRT) | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 3 months (T4), and 6 months (T5) postdischarge
  The Concise Health Risk Tracking (CHRT) is a 9-item survey that assesses suicidal thoughts and behaviors in the past week, with response options ranging 0-4. Total scores range 0-36, with higher scores indicating more severe suicidality.

SECONDARY OUTCOMES:
Change in Efficacy to Cope with Suicidal Thoughts and Urges Scale | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 3 months (T4), and 6 months (T5) postdischarge
  The Efficacy to Cope with Suicidal Thoughts and Urges Scale was designed to measure children's abilities to manage suicide-related thoughts and impulses. It contains 10 coping skills and children rate their confidence in their ability to use each coping skill to manage their suicidality. Responses range from 0 to 10 with 0 = Not at all confident, 5 = Somewhat confident, and 10 = Extremely confident.
Change in The Children's Hope Scale | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 3 months (T4), and 6 months (T5) postdischarge
  The Children's Hope Scale is a 6-item self-report measure of hope. Response options range from
  1 to 6, with 1 = None of the time and 6 = All of the time.
Change in My Thoughts About Therapy (MTT; REACH Framework Expectancy Scale) | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 3 months (T4), and 6 months (T5) postdischarge
  The MTT measures five factors of treatment engagement (Relationship, Expectancy, Attendance, Clarity, and Homework); the study will use the Expectancy scale only. Items are answered using a 4-point Likert-scale, with from 0 = "strongly disagree" and 3 = "strongly agree".
Change in Cunningham Treatment Engagement Readiness to Change Subscale | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 3 months (T4), and 6 months (T5) postdischarge
  The Cunningham Treatment Engagement Readiness to Change Subscale measures clients' level readiness to change with regard to treatment and behaviors. It contains 5 questions answered on a 5-point Likert-scale, from "strongly disagree" to "strongly agree".
Disposition change | Hospital discharge/approximately 72 hours after admission (T2)
  This is a dichotomous variable defined as discharge to home instead of inpatient psychiatric care and will be gathered from electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnna K Leyenaar, MD, PhD, MPH, Principal Investigator — Dartmouth Health
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded into the NIMH Data Archive (NDA).
  Data will be collected from approximately 109 adolescents 12-17 years of age. Measures include:
  1. Depression, Anxiety, and Stress Scale - Youth version (DASS-Y)
  2. Harkavy-Asnis Suicide Scale (HASS) - Suicide Attempt module
  3. Concise-Health Risk Tracking-Self Report (CHRT)
  4. Efficacy to Cope with Suicidal Thoughts and Urges Scale
  5. The Children's Hope Scale
  6. My Thoughts about Therapy Expectancy Scale
  7. Cunningham Treatment Engagement Readiness to Change Scale
  8. DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure for Youth
  9. RCADS-25 for Youth
Supporting Information: Study Protocol
Time Frame: All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: All those with access to the NDA will have access to our data.